CLINICAL TRIAL: NCT02177227
Title: Attune With TruMatch TM Personalized Solutions Instruments: A Prospective Randomized Controlled Trial Comparing Clinical and Economic Outcomes in Patients With a BMI Between 30 and 50
Brief Title: Attune With TruMatch TM Personalized Solutions Instruments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: DePuy Orthopaedics (Industry); Johnson & Johnson Medical Companies (Industry)
Responsible Party: Principal Investigator, Edward Vasarhelyi, Orthopaedic Surgeon, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Attune TruMatch
Record Dates: First submitted 2014-06-24; First posted 2014-06-27 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Obesity; Osteoarthritis
Keywords: Total Knee Arthroplasty (TKA); Attune; Primary Total Knee Prosthesis; TruMatch
MeSH Terms: conditions — Obesity; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Total Knee Arthroplasty with PSI (Experimental): Total Knee Replacement with the use of the Attune TruMatch (TM) Patient-Specific Instrumentation
  Interventions: Device: Attune TruMatch (TM) Patient-Specific Instrumentation
- Total Knee Replacement (No Intervention): Total Knee Replacement, as per Standard of Care

INTERVENTIONS:
Device: Attune TruMatch (TM) Patient-Specific Instrumentation — Patients to receive total knee replacement with TruMatch Patient-Specific Instrumentation
  Other Names: TruMatch Patient-Specific Instrumentation
  Arms: Total Knee Arthroplasty with PSI

SUMMARY:
The purpose of our study is to determine, using a prospective, randomized-controlled trial, the economic viability and clinical outcomes associated with patient-specific instrumentation (PSI) for total knee arthroplasty in an obese patient population.

DETAILED DESCRIPTION:
This is a randomized, blinded study. Following REB approval, eligible patients electing to undergo TKA will be identified by either the PI or co-investigators, and approached in an orthopaedic outpatient clinic to discuss enrolment into the study. Patients will be enrolled if they meet the prerequisite inclusion criteria and have signed an informed consent. Patients will then be randomized to undergo a TKA using PSI, or a conventional TKA. The randomization sequence will be computer generated using blocks of five. Preoperative Assessment At baseline, patients will complete a Knee Society Score (KSS), Short-Form 12 (SF-12) Questionnaire, and Western and McMaster University Osteoarthritis Index (WOMAC) questionnaire, and the European Quality of Life Scale Index (EQ-5D). The EQ-5D is a validated, reliable, and feasible outcome measure that provides a utility index. This utility index allows quality adjusted life years to be calculated following an intervention. The questionnaire is a 5-item standardized generic measure of health related quality of life that includes domains of mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. Each item is scored using a 3-point response scale and each combination of response choices describes a health state (resulting in 243 possible health states). Each health state can then be converted to a utility value ranging from 0 (worst) to 1.0 (best) using existing preference valuation data[22]. It has been valuated in both Canadian and American populations for use in assessing health-related quality of life [23, 24]. We will then calculate each patient's quality-adjusted life year (QALY). QALYs incorporate both length of life and quality of life into a single measure and are calculated by multiplying the utility value by the length of time spent in that health state. Additionally, a clinical assessment will be completed, including knee range of motion, ligamentous assessment, and evaluating for soft tissue contractures. Finally, patients will have 3-foot coronal and sagittal standing radiographs of their lower extremities at our institution. The standing mechanical axis of the involved limb will then be calculated. Skyline views will also be performed as part of the radiographic analysis. In order for appropriate preoperative planning, patients randomized to PSI will undergo a computed tomography (CT) scan of the surgical limb using the TruMatch TM scanning protocol. Following modifications made by the treating surgeon, the personalized patient instruments will be manufactured in standard fashion. Intraoperative Assessment On the day of surgery, patients will receive either a spinal or general anesthetic based on recommendations from an anesthetist, or personal preference. A non-sterile tourniquet will be applied to the operative limb. A mid-line skin incision followed by a medial parapatellar arthrotomy will be used for exposure. The femoral and tibial cuts will be made using conventional instrumentation in the control group, or the TruMatch TM Personalized Solutions Instruments in the treatment group. Soft tissue balancing, including releases and removal of osteophytes, will be performed at the discretion of the surgeon. The Attune TM components will be implanted using cement fixation. At the time of cementing the implants, patients will receive a parenteral weight-based dose of tranexamic acid (20 mg /kg), provided that there are no contra-indications. Prior to closure, patients will receive an intra-articular injection of an anesthetic cocktail. The parapatellar arthrotomy and subcutaneous tissue and skin will be closed in standard fashion. Post-operatively, patients will receive deep-vein thrombosis prophylaxis for 14-days post-operatively. They will also receive 24 hours of post-operative parenteral antibiotics. They will be assessed by physiotherapy, with weight-bearing and range of motion exercises beginning on post-operative day 0. Patients will be discharged from hospital once they have reached appropriate rehabilitative milestones outlined by our institution. Postoperative Assessment Patients will have routine follow-up with their surgeon at 2-, 6-, and 12-weeks, followed by 1-year and every other year thereafter. Three-foot coronal and full-length sagittal standing radiographs, as well as skyline views of the involved knee, will be taken at the 1-year postoperative visit. We will calculate the mechanical axis of the operative limb based on this postoperative radiographic assessment. The patients will complete the KSS, SF-12, WOMAC, and EQ-5D questionnaires at their 6-week, 12-week, and 1-year visits. These outcome questionnaires will be collected prospectively at 5-years and 10-years post-operatively through our institution's database. Assessors of both clinical outcomes and mechanical axis will be blinded to surgical intervention (conventional instrumentation versus PSI TKA). Patients will also receive a health care resource use diary to complete between follow-up intervals in order to collect outpatient direct and indirect costs associated with TKA. Costs Our institution's costs-accounting department will provide information regarding operating room costs, implant costs, and costs associated with routine care such as nursing, medications, and investigations. Physician-related costs will be acquired through Ontario Health Insurance Plan billing protocols. The outpatient cost analysis diary will capture direct, non-medical costs associated with TKA (see Appendix C). The data will be reported in Canadian dollars for the fiscal year in which the in-hospital cost data was derived. A sample database we are currently employing in an unrelated study can be provided if required. Cost-Utility Analysis Incremental Cost-Utility Ratio (ICUR) The ICUR represents the ratio of incremental cost to incremental utility. The incremental cost represents the additional cost of the PSI group compared to the conventional group. The costs will include all direct (operating room, hospital stay, rehabilitation, medications, investigations) and indirect costs (informal care, time lost to productivity). Similarly, the incremental utility is the mean difference in QALY between groups. Net Benefit Regression We will use the net benefit regression (NBR) framework to estimate the incremental net benefit (INB) of PSI [25]. An intervention is considered to be cost-effective if the INB is greater than zero. The net benefit regression method also provides a means to adjust for any potentially confounding factors and therefore allows greater statistical efficiency and provides a more precise estimate of the INB. We will include the following covariates in our regression models: baseline utility score, severity of osteoarthritis, age and number of comorbidities. To characterize the statistical uncertainty around our estimate of INB we will calculate 95% confidence intervals, and a cost-effectiveness acceptability curve (CEAC). Modeling To determine the cost-effectiveness of a new intervention, an economic decision model is appropriate when there are multiple existing sources of evidence to answer a question (e.g. randomized trials, cohort studies, registries, etc.) or to forecast the costs and/or outcomes beyond the follow-up period of the clinical trial. Given that PSI is a relatively new technology, there is no long-term data available to accurately determine the survival of the implant or the rate of revision. To accurately answer this question, we will prospectively follow the cohort long-term to determine survival rates of the implant.

ELIGIBILITY:
Inclusion Criteria:

* patients with body mass index (BMI; kg/m2) greater than 30 and less than or equal to 50
* Symptomatic knee osteoarthritis deemed most appropriately treated with total knee arthroplasty
* Patient greater than 19 and less than or equal to 70 years of age
* English-speaking

Exclusion Criteria:

* History of prior open knee surgery, infection, or previous knee trauma
* Simultaneous bilateral knee arthroplasty
* Underlying dementia, cognitive delay, any disorder, or geographic distance that would preclude the completion of the clinical questionnaires
* Inflammatory arthropathy
* Chronic pain syndrome
* Fibromyalgia

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Assessment of Possible Change in Radiographic Alignment | Pre-operatively, 6 weeks post-operatively, 1 year post-operatively
  Mechanical axis, sagittal alignment and tibial slope are to be assessed.

SECONDARY OUTCOMES:
Assessment of Possible Change in Peri-operative metrics | 1 year, 5 years and 10 years post-operatively
  Operating room time, hospital length of stay, complications and instances of re-admissions will be assessed.
Patient-completed questionnaires | pre-operatively, 6 weeks, 3 months, 1 year and then once each year.
  KSS WOMAC SF-12
Incremental cost-utility ratio | 1 year post-operatively, and each year until 10 years post-op
  Operating room time, hospital length of stay, complications and instance of readmission will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Edward M Vasarhelyi, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No